CLINICAL TRIAL: NCT03085394
Title: Preoperative Hexakapron Reduces Bleeding in Bariatric Surgery
Acronym: PHORBBS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment stopped, patients refuse to participate.
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, David Goitein MD, Head, Bariatric and Metabolic Surgery, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMC-17-3846
Record Dates: First submitted 2017-03-19; First posted 2017-03-21 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Intra-Operative Injury - Other; Post Operative Hemorrhage; Tranexamic Acid
Keywords: Morbid Obesity; Sleeve gastrectomy
MeSH Terms: conditions — Postoperative Hemorrhage; Obesity, Morbid | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Active Comparator): Preoperative intravenous administration of 2g tranexamic acid in 10ml fluid.
  Interventions: Drug: tranexamic acid
- Control Arm (Placebo Comparator): Preoperative intravenous administration of 10ml normal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tranexamic acid — Preoperative intravenous administration of 2 grams tranexamic acid in 10 ml saline
  Other Names: Hexakapron
  Arms: Treatment arm
Drug: Placebo — Preoperative intravenous administration of 10 ml saline
  Arms: Control Arm

SUMMARY:
Prophylactic use of tranexamic acid to reduce intra and postoperative bleeding in primary sleeve gastrectomy procedures will be studied.

DETAILED DESCRIPTION:
Patients scheduled for primary laparoscopic sleeve gastrectomy for the treatment of morbid obesity will be assigned to receive tranexamic acid vs. placebo before surgery. Intraoperative bleeding will be scored, as well as postoperative bleeding and blood or blood-product requirements. POstoperative venous thromboembolic events will be recorded up to 2 months following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity
* Approved and scheduled for laparoscopic sleeve gastrectomy

Exclusion Criteria:

* Previous bariatric surgery
* Platelet count under 100,000
* Concurrent anticoagulation treatment
* Previous venous/atrerial thromboembolic event
* Known allergy to tranexamic acid
* History of heparin induced thrombocytopenia
* Oral contraceptive use
* Female hormonal replacement therapy
* Active thromboembolic state
* Genetic hypercoagulable state

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Treatment efficiency (lowering/preventing clinically significant bleeding) | 1 week
  The efficiency of preoperative tranexamic acid administration in lowering/preventing clinically significant bleeding.
Treatment safety (administering tranexamic acid preoperatively without promoting thromboembolic events) | 2 months
  The safety of administering tranexamic acid preoperatively without promoting thromboembolic events

SECONDARY OUTCOMES:
Need for reintervention | 1 week
  The proportion of patients requiring invasive intervention (percutaneous/operative) due to bleeding
Procedure change | 1 day
  The proportion of patients requiring alteration of intended procedure due to bleeding.
Blood/blood product requirement | 1 week
  The usage of blood/blood products after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel